CLINICAL TRIAL: NCT02974023
Title: Efficacy of "Pain Gear" in Patients With Chronic Musculoskeletal Pain
Status: Withdrawn | Type: Observational
Why Stopped: Study not started due to the Regulatory and administrative issues of Universities in Vietnam
Sponsor: PharmEvo Pvt Ltd (Industry)
Collaborators: BioElectronics Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: PE/PAINGEAR/09/2016
Record Dates: First submitted 2016-11-22; First posted 2016-11-28 (Estimated); Last update posted 2018-10-03 (Actual); Status verified 2016-12

CONDITIONS: Chronic Musculoskeletal Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Pain Gear — PainGear [ActiPatch®] (BioElectronics Corporation, MD, USA) has been recently introduced as an 'topical' analgesic for localized musculoskeletal pain. PainGear is a noninvasive, low power, easy to use, pulsed shortwave therapy device for localized musculo¬skeletal pain.
  Other Names: ActiPatch

SUMMARY:
The current study was designed to evaluate the effectiveness and safety of the device in the common areas of the body affected by different causes of musculoskeletal pain in Vietnamese population in real life situation.

DETAILED DESCRIPTION:
PainGear [ActiPatch®] (BioElectronics Corporation, MD, USA) has been recently introduced as an 'topical' analgesic for localized musculoskeletal pain. PainGear is a noninvasive, low power, easy to use, pulsed shortwave therapy device for localized musculoskeletal pain. The device does not produce heat or any sensation. There are two basic requirements to use the device, switching it on via an on/off switch, and affixing the device over the target area of the body. The area of treatment is confined to the area within the 11.5-cm diameter loop antenna covering an area of 100 cm2, the antennae is circular, soft and flexible and can be shaped to fit the area/location being treated as required. The device can be used up to 24 h per day and is placed over the area of localized pain either using medical tape or a specifically designed wrap.

In a randomized, double-blind, placebo-controlled clinical trial, patients with radiographic evidence of knee OA (osteoarthritis) and persistent pain higher than 40mm on the visual analog scale (VAS) were recruited. The trial consisted of 12 h daily treatment for 1 month in 60 knee OA patients. After 1 month, PainGear induced a significant reduction in VAS pain and Western Ontario and McMaster Universities Arthritis Index (WOMAC) scores compared with placebo. Additionally, pain tolerance and physical health improved in PainGear -treated patients. Twenty-six per cent of patients in the PainGear group stopped NSAID/analgesic therapy. No adverse events were detected.

ELIGIBILITY:
Inclusion Criteria:

* Chronic musculoskeletal pain of more than 6 month duration
* Participant is willing and able to give informed consent for participation in the trial.
* In the Investigator's opinion, is able and willing to comply with all trial requirements.
* Male or female ages 18-80 years old
* A current VAS pain rating ≥5/10
* Able to complete and tolerate treatment for the study period.

Exclusion Criteria:

* Pregnant Woman
* Current implanted cardiac demand pacemakers, defibrillators, cardiac pumps, spinal stimulators or other implanted electronic devices.
* Patients using personal home based electrical stimulation devices
* Active psychiatric disorders (as evidenced by use of antipsychotic or medication).
* Patients diagnosed with history of significant mood disorder will be excluded (depression or anxiety with adequate control would be acceptable).
* Scheduled elective surgery or other procedures requiring general anesthesia during the trial.
* Participant with life expectancy of less than 6 months, or inappropriate for placebo medication.
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial.
* Participants who are not able to understand verbal or written English, and for whom adequate translation/interpretation cannot be readily obtained

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from Low back pain and arthritis.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-06-30 (Actual); Primary Completion 2017-10-30 (Actual); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
To assess difference in subjective pain with the use of PainGear for 2 weeks. | 2 weeks
  [ Time Frame: Change from baseline visual analogue score over the course of 2 weeks]

SECONDARY OUTCOMES:
To record change in frequency of other analgesic modalities utilization | 2 weeks period
  [ Time Frame: Change from baseline analgesic modalities usage over the course of 2 weeks period, to be recorded in modalities chart]
To assess difference in Pain-related disability, indexed by the Oswestry Disability Index (ODI) | 2 weeks, recorded on 1st and 14th day
  [ Time Frame: Change from baseline ODI score at 2 weeks, recorded on 1st and 14th day ]
To assess patients satisfaction with two weeks therapy of PainGear | 14th day
  [Time Frame: 14th day]